CLINICAL TRIAL: NCT02889380
Title: A Retrospective Study in Chinese Good Prognosis Patients Undergoing ART Treatment to Investigate the Factors Associated With the Pregnancy Outcome of GnRH Antagonist IVF/ICSI Cycles
Brief Title: A Retrospective Study in Chinese Good Prognosis Patients Undergoing Assisted Reproductive Technology (ART) Treatment
Acronym: FASSION
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: MS200106-0004
Record Dates: First submitted 2016-08-30; First posted 2016-09-05 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Infertility
Keywords: Infertility; Cetrotide; Assisted reproductive technology (ART)
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cetrotide: This study will retrospectively collect the data from the subjects who had been treated with 0.25 milligram (mg) of Cetrotide injection daily in a fixed or flexible antagonist protocol with an available assisted reproductive technology (ART) outcome.
  Interventions: Drug: No Intervention

INTERVENTIONS:
Drug: No Intervention — This study will retrospectively collect the data from the subjects who had been treated with 0.25 mg of Cetrotide injection daily in a fixed or flexible antagonist protocol with an available ART outcome.

SUMMARY:
This is a multicenter retrospective study in good prognosis Chinese patients. Data will be collected from infertile women who underwent first in vitro fertilization (IVF)/intra cytoplasmic sperm injection (ICSI) using a Gonadotropin releasing hormone (GnRH) antagonist (Cetrotide) protocol at about 4 IVF centers to investigate the factors associated with clinical pregnancy rate. The definition of the good prognosis subjects is, age not more than 35 years old, Baseline serum Follicle-stimulating hormone (FSH) level no more than 10 milliinternational units (mIU)/milliliter (ml), Body mass index (BMI) not more than 30 kilogram per meter square (kg/m^2), previously underwent no more than 3 IVF/ICSI cycles, and the total dose of Gonadotropin used no more than 2500 IU in current cycle. No intervention(s) will be administered on the subjects. Data required to investigate the factors associated with the pregnancy outcome of GnRH antagonist IVF cycle will be collected from the subjects' medical records into database through electronic data capture system and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women who underwent the first GnRH antagonist IVF/ICSI-ET (Embryo Transfer) cycle with an available ART outcome
* Used Cetrotide in a fixed or flexible antagonist protocol
* Age not more than 35 years old
* Baseline serum Follicle-stimulating hormone (FSH) level not more than 10 milliinternational unit per milliliter (mIU/ml)
* Body mass index (BMI) not more than 30 kilogram per meter square (kg/m^2)
* Normal uterine cavity

Exclusion Criteria:

* Previously underwent 3 or more IVF/ICSI cycles
* The total dose of Gonadotropin used was more than 2500 IU in current cycle
* Administration of daily 0.125 milligram (mg) Cetrotide
* Received an agonist trigger
* Use of clomiphene citrate or letrozole during cycles
* Presence of endometriosis Grade 3 to 4, confirmed or suspected
* Presence of uni-or-bilateral hydrosalpinx
* Known history of recurrent miscarriages

Max Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Infertile Chinese women who underwent the first Gonadotropin releasing hormone (GnRH) antagonist in vitro fertilization (IVF)/intra cytoplasmic sperm injection - Embryo Transfer (ICSI-ET) cycle with an available assisted reproductive technology (ART) outcome.
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2017-04-26 (Actual); Study Completion 2017-04-26 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate | 5 months
  Number of clinical pregnancies expressed per 100 initiated cycles, aspiration cycles, and embryo transfer cycles. Initiated cycle: an assisted reproductive technology (ART) cycle in which the woman receives specific medication for ovarian stimulation, or monitoring in the case of natural cycles, with the intention to treat, irrespective of whether or not follicular aspiration is attempted. Aspiration cycle Initiated ART cycle in which one or more follicles are punctured and aspirated irrespective of whether or not oocytes are retrieved. Embryo transfer cycle: an ART cycle in which one or more embryos are transferred into the uterus or fallopian tube.
Implantation Rate | 5 months
  Implantation rate = (The number of gestational sacs observed divided by the number of embryos transferred)*100
Ongoing Pregnancy Rate | 5 months
  Ongoing pregnancy rate per embryo transfer cycles = (Number of Ongoing pregnancy/Number of embryo transfer cycles)*100 and ongoing pregnancy rate per initiated cycles = (Number of Ongoing pregnancy/Number of initiated cycles) *100
Incidence and Severity of Ovarian Hyperstimulation Syndrome (OHSS) | 5 months
Cycle Cancelled Rate | 5 months
  Cycle cancelled rate = (Number of subjects with terminated in vitro fertilization (IVF) or intra cytoplasmic sperm injection (ICSI) treatment/Number of initiated cycles)*100
Early Miscarriage Rate | 5 months
  (Number of Early miscarriages/Number of clinical pregnancies)*100
Live Birth Rate | 5 months
  Number of live births expressed per 100 initiated cycles, aspiration cycles or embryo transfer cycles. When delivery rates are given, the denominator (initiated, aspirated, or embryo transfer cycles) will be specified
Type of Gonadoptropin | 5 months
Brand of Gonadotropin | 5 months
Total Dose of Gonadotropin | 5 months
Duration of Gonadotropin Administration | 5 months
Cetrotide Start Day | up to 5 months
Leading Follicle Size on the Day of Starting Cetrotide | on the day of starting Cetrotide (up to 5 months)
Serum Luteinizing Hormone (LH) Level on the Day of Starting Cetrotide | on the day of starting Cetrotide (up to 5 months)
Serum Estradiol (E2) Level on the Day of Starting Cetrotide | on the day of starting Cetrotide (up to 5 months)
Serum Luteinizing Hormone (LH), Level on the Day of Human Chorionic Gonadotropin (hCG) Triggering | 5 months
Serum Estradiol (E2) Level on the Day of Human Chorionic Gonadotropin (hCG) Triggering | on the day of hCG triggering (up to 5 months)
Progesterone Level on the Day of Human Chorionic Gonadotropin (hCG) Triggering | on the day of hCG triggering (up to 5 months)
Number of Follicles With Size 14 milimeter (mm) or More on the Day of Human Chorionic Gonadotropin (hCG) Triggering | on the day of hCG triggering (up to 5 months)
Endometrial Thickness on the Day of Human Chorionic Gonadotropin (hCG) Triggering | on the day of hCG triggering (up to 5 months)
Serum Luteinizing Hormone (LH) Level on the Day of Observed Premature Luteinizing Hormone (LH) Rise | on the day of observed premature LH rise (up to 5 months)
  Subjects will be characterized as having a premature LH rise if any measured LH value during follicular recruitment will more than (>) 10 International Units Per Litre (IU/L) up to and including the day of the trigger
Serum Estradiol (E2) Level on the Day of Observed Premature Luteinizing Hormone (LH) Rise | on the day of observed premature LH rise (up to 5 months)
  Subjects will be characterized as having a premature LH rise if any measured LH value during follicular recruitment will more than (>) 10 International Units Per Litre (IU/L) up to and including the day of the trigger
Serum Progesterone Level on the Day of Observed Premature Luteinizing Hormone (LH) Rise | on the day of observed premature LH rise (up to 5 months)
  Subjects will be characterized as having a premature LH rise if any measured LH value during follicular recruitment will more than (>) 10 International Units Per Litre (IU/L) up to and including the day of the trigger
Number of Follicles With Size 14 mm or More on the Day of Observed Premature Luteinizing Hormone (LH) Rise | on the day of observed premature LH rise (up to 5 months)
  Subjects will be characterized as having a premature LH rise if any measured LH value during follicular recruitment will more than (>) 10 International Units Per Litre (IU/L) up to and including the day of the trigger
Endometrial Thickness on the Day of Observed Premature Luteinizing Hormone (LH) Rise | on the day of observed premature LH rise (up to 5 months)
  Subjects will be characterized as having a premature LH rise if any measured LH value during follicular recruitment will more than (>) 10 International Units Per Litre (IU/L) up to and including the day of the trigger
Serum Progesterone Level on the Day of Observed Premature Progesterone Rise | on the day of observed premature progesterone rise (up to 5 months)
  Premature progesterone rise: A rise in serum progesterone levels above 1.5 nanogram/milliliter (ng/ml) towards the end of the follicular phase up to and including the day of the trigger
Number of Oocytes Obtained | 5 months
Number of Mature Metaphase II Oocytes Obtained | 5 months
Fertilization Rate | 5 months
Total Number of Embryos on Day 3/Blastocysts on Day 5 | Day 3 and Day 5
Number of Cryopreservation Embryos/Blastocysts on Day 3 or Day 5 | Day 3, Day 5
Number of Embryos/Blastocysts Transferred on Day 3 or Day 5 | Day 3, Day 5
Number of Good Quality Embryos/Blastocysts Transferred | up to 5 months
Age | Baseline
Duration of Infertility | Baseline
Type of Infertility | Baseline
Body Mass Index (BMI) | Baseline
Smoking Status | Baseline
Cause of Infertility | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono Co., Ltd., China
Locations (4):
- China (4):
  - Peking University Third Hospital, Beijing
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Reproductive Hospital Affiliated to Shandong University, Shandong
  - Reproductive & Genetic hospital of CITIC-XIANGYA, Xiangya